CLINICAL TRIAL: NCT02916056
Title: Open Label Extension Study for Continued Safety and Efficacy Evaluation of Azeliragon in Patients With Mild Alzheimer's Disease
Brief Title: 2-Year Extension Study of Azeliragon in Subjects With Alzheimer's Disease (STEADFAST Extension)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not due to safety but due to a lack of efficacy at the 5 mg azeliragon dose.
Sponsor: vTv Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTP488-303
Record Dates: First submitted 2016-08-10; First posted 2016-09-27 (Estimated); Results first posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; RAGE; ADAS-cog; CDR-sb
MeSH Terms: conditions — Alzheimer Disease | interventions — azeliragon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azeliragon 5 mg (Experimental): Azeliragon (TTP488) 5mg orally once daily for 2 years
  Interventions: Drug: Azeliragon 5mg

INTERVENTIONS:
Drug: Azeliragon 5mg
  Other Names: TTP488

SUMMARY:
This is an open-label extension study in patients with mild Alzheimer's disease who have completed participation in the azeliragon Phase 3 (STEADFAST) trial. Patients will receive azeliragon 5 mg/day for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of Study TTP488-301 through the Month 18 Visit without ongoing serious adverse events or history of serious adverse drug reactions during study TTP488-301.
* Patients must enroll in the present study within 7 days of completion of study TTP488-301.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally authorized representative) and caregiver/informant has been informed of all pertinent aspects of the study. Participants must be able to provide assent (where this is in accordance with local laws, regulations and ethics committee policy) and assent may be re-evaluated during the study at regular intervals.
* Participants and caregiver/informants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* The subject must have a reliable caregiver/informant with regular contact (i.e., 10 hours a week as combination of face-to-face visits and telephone contact acceptable) who will facilitate the subject's full participation in the study. Caregivers/informant must have sufficient subject interaction to be able to provide meaningful input into the rating scales administered in this study where caregiver/informant input is required, in particular the CDR and evidence of this should be documented in source documentation. Participants who reside in assisted living facilities are permitted provided that they meet caregiver/informant criteria.
* Participants and caregiver/informants must be able to read, write, and speak the language in which psychometric tests are provided with visual and auditory acuity (corrected) sufficient to allow for accurate psychometric testing.
* Subject must be able to ingest oral medications.

Exclusion Criteria:

* The subject is felt by the investigator to be unsuitable (on the basis of health, compliance, caregiver availability, or for any other reason) for inclusion in the study.
* Subjects with serious suicide risk. If there are "yes" answers on items 4, 5 or on any behavioral question of the C-SSRS, a suicide risk assessment must be done by a qualified mental health professional with expertise in the evaluation of suicidality in the elderly (e.g., psychiatrist, geriatrician or neurologist specializing in treatment of patients with AD) to determine whether it is safe for the subject to participate in the study.
* Subjects demonstrating a QTcF > 480 msec or a >45 msec change from the TTP488-301 Baseline value based on the locally read ECG performed at the TTP488-301 Month 18 Visit (TTP488-303 Baseline). Participants with known history of bundle branch block (either right or left) are allowed if absolute QTcF value does not exceed 500 msec. Participants with a functioning pacemaker, indicated by an ECG displaying paced rhythm, are allowed with no QTc upper limit.
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may prevent the subject from completing the 2-year study or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Gooch, Ph.D., Study Director — vTv Therapeutics LLC
Locations (65):
- United States (59):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Bellflower, California
  - Costa Mesa, California
  - Fullerton, California
  - Glendale, California
  - Imperial, California
  - Irvine, California
  - Laguna Hills, California
  - Long Beach, California
  - Riverside, California
  - San Bernardino, California
  - Santa Ana, California
  - Atlantis, Florida
  - Delray Beach, Florida
  - Hallandale, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Lake Worth, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Miami Lakes, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Sunrise, Florida
  - The Villages, Florida
  - Columbus, Georgia
  - Chicago, Illinois
  - Fairway, Kansas
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Newton, Massachusetts
  - Plymouth, Massachusetts
  - Quincy, Massachusetts
  - Hattiesburg, Mississippi
  - Creve Coeur, Missouri
  - St Louis, Missouri
  - Princeton, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Lake Success, New York
  - New York, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Shaker Heights, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Plains, Pennsylvania
  - East Providence, Rhode Island
  - Cordova, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Wichita Falls, Texas
  - Murray, Utah
  - Kirkland, Washington
- Canada (6):
  - Calgary, Alberta
  - Medicine Hat, Alberta
  - Chatham, Ontario
  - Toronto, Ontario
  - Gatineau, Quebec
  - Greenfield Park, Quebec

REFERENCES:
- See also: Related Info — http://www.livingsteadfast.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants who completed TTP488-301 were enrolled into the TTP488-303 Open label extension from December 2016 through April 2018 in the United States and Canada.
Groups:
- Azeliragon 5 mg: Azeliragon (TTP488) 5mg orally once daily
Period: Overall Study
Arm/Group | Azeliragon 5 mg
Started | 297
Completed | 0
Not Completed | 297
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 1
Not completed — Other | 12
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 8
Not completed — Study Terminated by Sponsor | 269

BASELINE CHARACTERISTICS:
Arm/Group | Azeliragon 5 mg
Number analyzed (Participants) | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.9 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144
  Male | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31
  Not Hispanic or Latino | 266
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 9
  White | 280
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Treatment-Emergent Adverse Event
Time Frame: up to 18 months
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Azeliragon 5 mg
Number analyzed (Participants) | 297
Participants | 193

ADVERSE EVENTS:
Time Frame: Adverse events were collected from consent through end of study participation. Duration of study participation was up to 456 days.
Arm/Group | Azeliragon 5 mg
All-Cause Mortality (participants affected / at risk) | 0/297
Serious Adverse Events (participants affected / at risk) | 25/297
Other Adverse Events (participants affected / at risk) | 137/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azeliragon 5 mg (N=297)
Transient ischaemic attack (Nervous system disorders) | 3
Ataxia (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Complex partial seizures (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Bacterial prostatitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Orthostatic hypotension (Vascular disorders) | 2
Aortic stenosis (Vascular disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azeliragon 5 mg (N=297)
Dizziness (Nervous system disorders) | 12
Headache (Nervous system disorders) | 7
Upper respiratory tract infection (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 9
Depression (Psychiatric disorders) | 13
Insomnia (Psychiatric disorders) | 8
Fall (Injury, poisoning and procedural complications) | 29
Laceration (Injury, poisoning and procedural complications) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Fatigue (General disorders) | 7
Gait disturbance (General disorders) | 7
Weight decreased (Investigations) | 9
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Where PI requires the use of the Study Results for publication, the PI shall seek the Sponsor's written approval which shall not be unreasonably withheld; provided, however, that (i) Sponsor may require removal of any Confidential Information of Sponsor or may delay publication for a reasonable period of time in order to secure protection any IP Rights; and, (ii) as the Study is designed as a multi-center Study, no publication shall be made until after the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT02916056/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT02916056/SAP_001.pdf